CLINICAL TRIAL: NCT05267457
Title: Associations of Plasma Vanadium Concentrations With Gestational Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Liegang Liu (Other)
Responsible Party: Sponsor-Investigator, Liegang Liu, Professor, Huazhong University of Science and Technology
Organization: Huazhong University of Science and Technology (Other)
Other Study IDs: XQL202202
Record Dates: First submitted 2022-02-24; First posted 2022-03-04 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Gestational Diabetes
Keywords: Vanadium; Gestational diabetes mellitus
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Gestational diabetes mellitus: Gestational diabetes mellitus (GDM) was diagnosed according to the American Diabetes Association criteria, which is based on the "one-step" approach recommended by the International Association of Diabetes and Pregnancy Study Groups. All women underwent a 75g OGTT in the morning after an overnight fast, with plasma glucose measurement fasting and at 1 and 2 hours. The criteria for GDM diagnosis was to have at least one abnormal value: Fasting glucose ≥ 5.1 mmol/L (92 mg/dL), 1 h glucose ≥ 10.0 mmol/L (180 mg/dL), 2 h glucose ≥ 8.5 mmol/L (153 mg/dL).
  Interventions: Other: Plasma vanadium concentration
- Healthy pregnant women: Pregnant women with fasting glucose < 5.1 mmol/L (92 mg/dL), 1 h glucose < 10.0 mmol/L (180 mg/dL) and 2 h glucose < 8.5 mmol/L (153 mg/dL) were considered as healthy controls. Controls were randomly selected and individually matched to cases by age (± 2 years), gestational age (± 2 weeks) and parity.
  Interventions: Other: Plasma vanadium concentration

INTERVENTIONS:
Other: Plasma vanadium concentration — Plasma vanadium concentrations were measured using inductively coupled plasma mass spectrometry (ICP-MS) (Agilent 7700 Series, United States)

SUMMARY:
Background: Vanadium compounds have been shown to exert insulin-mimetic effects and thereby control glucose homeostasis. However, studies regarding the levels of vanadium and gestational diabetes mellitus (GDM) are limited and have inconsistent outcomes.

Objective: The aim of this study was to investigate the association of plasma vanadium concentrations with gestational diabetes mellitus (GDM).

Design: A hospital-based case-control study was carried out in urban Wuhan, China from August 2012 to April 2015. Pregnant women who screened for GDM at the outpatient clinics of the Department of Endocrinology, Tongji Hospital were invited to participant in the study. The inclusion criteria were as follows: 1) age ≥ 20 and ≤ 43 years; 2) gestational age at GDM screening ≥ 24 weeks; 3) singleton pregnancy. The investigators excluded women who met any of the following items: history of diabetes (including but not limited to GDM), cardiovascular disease, cancer or other systemic diseases; pharmacologic treatment or dietary supplement use that might influence glucose or lipids metabolism; accompanied by other pregnancy complications; incomplete basic information. The diagnosis of GDM can be made if one or more glucose values are above the cut points of 5.1, 10.0 and 8.5 mmol/L at fasting, 1 and 2 h during a 75-gram oral glucose tolerance test (OGTT). Controls were randomly selected and individually matched to cases by age (± 2 years), gestational age (± 2 weeks) and parity. Finally, 252 GDM cases and 252 matched controls were selected in this study. All participants gave written informed consent before enrolling in the study. Fasting blood samples (≥ 8 h overnight fasting) were collected using anticoagulant tubes and centrifuged at 3000 rpm for 5 min. Plasma were separated from blood cells and stored at -80 ℃ for further assay. Plasma vanadium concentrations were measured using inductively coupled plasma mass spectrometry. Conditional logistic regression and restricted cubic spline model were used to evaluate the associations between plasma vanadium and odds of GDM.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 20 and ≤ 43 years;
* Gestational age at GDM screening ≥ 24 weeks;
* Singleton pregnancy;

Exclusion Criteria:

* History of diabetes (including but not limited to GDM), cardiovascular disease, cancer or other systemic diseases;
* History of receiving pharmacological treatment known to affect glucose metabolism;
* Incomplete basic information.

Ages: 20 Years to 43 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All the participants enrolled were Chinese women. They gave informed written consent to the study and did not take any medication known to affect glucose tolerance or insulin secretion before participation.
Sampling Method: Probability Sample
Enrollment: 504 (Actual)
Dates: Start 2012-08-01 (Actual); Primary Completion 2015-04-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Gestational diabetes mellitus | From August 2012 to April 2015
  Glucose intolerance with onset or first diagnosis during pregnancy. The diagnosis of GDM can be made if one or more glucose values are above the cut points of 5.1, 10.0 and 8.5 mmol/L at fasting, 1 and 2 h during a 75-gram oral glucose tolerance test.